CLINICAL TRIAL: NCT02875626
Title: Role of Indocyanine Green (ICG) for Detection of Sentinel Nodes in Breast Cancer (FLUO-BREAST)
Brief Title: Role of Indocyanine Green (ICG) for Detection of Sentinel Nodes in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association Pour La Recherche des Thérapeutiques Innovantes en Cancérologie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FLUOBREAST
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Infracyanine green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Infracyanine (Experimental): In the beginning of the intervention, a periareolar injection of the Infracyanine will be carried out (Infracyanine®, 2ml to 2.5mg/ml whether 3.2nM).
  Interventions: Drug: Infracyanine

INTERVENTIONS:
Drug: Infracyanine — In the beginning of the intervention, a periareolar injection of the Infracyanine will be carried out (Infracyanine®, 2ml to 2.5mg/ml whether 3.2nM).
  Other Names: indocyanin green

SUMMARY:
This is a single-center prospective study evaluating the diagnostic performance and safety of Infracyanine in women with early breast cancer whose the research of sentinel node(s) combines isotopes and Infracyanine.

DETAILED DESCRIPTION:
Visits:

Screening:

Complete physical and gynecological examination by surgical oncologist Informed and signed consent form. The intervention will be planned within one month.

Intervention:

In the beginning of the intervention, a periareolar injection of the Infracyanine will be carried out (Infracyanine®, 2ml to 2.5mg/ml whether 3.2nM).

The search or sentinel node will be made using a infrared camera for transcutaneous visualization Secondly, data lymphoscintigraphy may be communicated to the surgeon. The nodes are identified as SN fluorescent nodes and / or radioactive nodes.

* All radioactive nodes and / or fluorescent will be deleted
* Reports of anatomy fluorescent SN and / or hot

Next visit:

The patient will be reviewed in consultation in the months following the itervention for a clinical examination, the collection of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Female age > 18 years
2. Invasive breast cancer ≤ 5 cm, unifocal bifocal or multifocal
3. Diagnosis confirmed by biopsy
4. Breast cancer extended in situ
5. First surgical treatment

Exclusion Criteria:

1. Neoadjuvant chemotherapy or hormone therapy.
2. Multicentric tumor
3. Pregnant patient
4. Ongoing participation in another clinical trial with an investigational drug

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-09; Primary Completion 2019-02 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the SN detection rate during surgery by fluorescence, by isotopes, by combining the two. The detection rate is defined by the number of patient | During surgery
  The detection rate is defined by the number of patient who at least one axillary sentinel node detected by fluorescence and / or isotope intraoperatively / number of female patients injected.

SECONDARY OUTCOMES:
The time between the incision and removal of the first sentinel node identified | During surgery
The sensitivity of indocyanine green compared to the technical reference ( percentage of nodes detected by the isotope and which are also detected by the indocyanine green ) | During surgery
The wrong negative rate (number of female patients in whom at least one metastatic sentinel node has been detected by isotope and not by ICG) | During surgery
Technical direct cost | during the study
Incidence rates of allergic reactions | From screening till 1 month after the surgery
Severity of allergic reactions (grade 1 to 5 according to Ring and al 38 ) | From screening till 1 month after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte NGO, MD, Principal Investigator — Hôpital Européen Georges-Pompidou
Locations (1):
- Hôpital Européen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ngo C, Sharifzadehgan S, Lecurieux-Lafayette C, Belhouari H, Rousseau D, Bonsang-Kitzis H, Crouillebois L, Balaya V, Oudard S, Lecuru F, Elaidi RT. Indocyanine green for sentinel lymph node detection in early breast cancer: Prospective evaluation of detection rate and toxicity-The FLUOBREAST trial. Breast J. 2020 Dec;26(12):2357-2363. doi: 10.1111/tbj.14100. Epub 2020 Oct 22. PMID 33094498